CLINICAL TRIAL: NCT07329894
Title: A Single-center, Non-randomized, Open-label Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Efficacy of XH001 Injection Combined With Neoantigen Vaccine-induced Tumor-specific T-cell Injection in Advanced Gastrointestinal Cancer
Brief Title: Safety, Tolerance and Preliminary Efficacy of XH001 Injection Combined With Neoantigen Vaccine-induced Tumor-specific T-cell Injection in Advanced Gastrointestinal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Collaborators: NeoCura (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XKY-C-007
Record Dates: First submitted 2025-12-11; First posted 2026-01-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Cancer
Keywords: Tumor Neoantigen Vaccine; Gastrointestinal Cancer; Adoptive Cell Therapy
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tumor neoantigen vaccine and tumor vaccine-induced specific T-cell Arm 1 (Experimental): Tumor neoantigen vaccine; Tumor vaccine-induced specific T-cell Dose 1
  Interventions: Drug: XH001 injection; Drug: Tumor vaccine-induced specific T-cell injection
- Tumor neoantigen vaccine and tumor vaccine induced specific T-cell Arm 2 (Experimental): Tumor neoantigen vaccine; Tumor vaccine induced specific T-cell dose 2
  Interventions: Drug: XH001 injection; Drug: Tumor vaccine-induced specific T-cell injection

INTERVENTIONS:
Drug: XH001 injection — mRNA tumor neoantigen vaccine
Drug: Tumor vaccine-induced specific T-cell injection — Adoptive T Cell Therapy

SUMMARY:
The goal of this clinical trial is to learn the safety of tumor neoantigen vaccine combined with neoantigen vaccine induced T-cell in treating advanced gastrointestinal cancer in adults. It will also learn if the combined treatment works to treat advanced gastrointestinal cancer.The main questions it aims to answer are:What medical problems do participants have when using the combined treatment? Does tumor neoantigen vaccine combined with neoantigen vaccine induced T-cell eliminate or shrink the tumor, and can it prolong the patient's survival period?

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Aged between 18 and 70 years old, male or female.
* Advanced gastrointestinal cancer that has been diagnosed by histological and/or cellular pathology, and which has failed to respond to second-line standard treatment or is intolerant to it, or is not suitable for standard treatment at this stage.
* According to the RECIST 1.1 criteria for evaluating the efficacy of solid tumors, there must be at least one measurable lesion as the target lesion for efficacy evaluation. The total diameter of the overall tumor lesion (excluding bone metastases) should be ≤ 100mm, and the diameter of a single tumor lesion should be ≤ 30mm. If the lesion that has received local treatment (radiotherapy, ablation, vascular intervention, etc.) is the only lesion, then there must be clear imaging evidence of disease progression for this lesion.
* Expected survival duration ≥ 12 weeks.
* Adequate organ and bone marrow function.

Exclusion Criteria:

* Requires long-term systemic administration of antiallergic drugs, or has severe hypersensitivity reactions (≥Grade 3) to XH001 injection and/or any of its excipients.
* Central nervous system metastases with symptoms, and/or meningeal metastases.
* Having received immunomodulatory drug therapy within 2 weeks prior to the first administration day (D1) of XH001 injection.
* Suffer from skin diseases that may prevent the intradermal injection from reaching the target area (such as psoriasis).
* Subjects with toxic side effects from previous treatment that have not recovered to CTCAE grade≤2, excluding hair loss.
* Subjects who received systemic steroid treatment (daily dose exceeding 10mg of prednisone equivalent) or any other form of immunosuppressive treatment within 7 days before the first administration of XH001 injection, excluding:1) Intranasal inhalation of local steroids or local steroid injection (such as intra-articular injection); 2) Systemic corticosteroid treatment not exceeding 10mg/day of prednisone or its equivalent physiological dose.
* Subjects who have previously received therapeutic tumor vaccines or therapeutic cell therapy products.
* Previously received allogeneic hematopoietic stem cell or allogeneic bone marrow transplantation, or previously received solid organ transplantation, or currently using immunosuppressive drugs.
* Have active or poorly controlled severe infections during screening period.
* Virological tests show positive for human immunodeficiency virus antibodies, hepatitis B surface antigen and/or hepatitis B core antibody with hepatitis B virus DNA > 1000 IU/ml, positive for hepatitis C virus antibodies, and positive for Treponema pallidum specific antibodies.
* Patients with other malignancies within 5 years before enrollment, except for those with a history of appropriately treated and cured cervical carcinoma in situ, breast carcinoma in situ, or skin basal cell carcinoma.
* Any history of autoimmune diseases.
* Known to have active pulmonary tuberculosis (TB).
* Patients who have received systemic chemotherapy, radiotherapy, molecular targeted therapy, biological immunotherapy, hormone therapy or unapproved clinical trial drugs/instruments within 2 weeks before screening.
* Subjects who are still participating in other clinical trials during the screening period.
* Pregnant or lactating women.
* Other severe, acute, or chronic medical or psychiatric conditions, or laboratory abnormalities, that, to the investigator's discretion, may increase the risks of participating in the trial or may interfere with the interpretation of the trial results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Adverse event | 12 months
  Incidence and severity of adverse events as assessed by Common Terminology Criteria for Adverse Events [CTCAE] V5.0
Dose Limiting Toxicity | From reinfusion of neoantigen vaccine-induced tumor-specific T cells to 28 days after the reinfusion
  Safety events occurring within 28 days after the reinfusion of neoantigen vaccine-induced tumor-specific T cells and related to this cell therapy.

SECONDARY OUTCOMES:
ORR | 24 months
  Objective Response Rate
PFS | 24 months
  Progression-Free Survival
DCR | 24 months
  Disease Control Rate
OS | 36 months
  Overall Survival
BOR | 24 months
  Best Overall Response
DOR | 24 months
  Duration of Response

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Gobroad Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rojas LA, Sethna Z, Soares KC, Olcese C, Pang N, Patterson E, Lihm J, Ceglia N, Guasp P, Chu A, Yu R, Chandra AK, Waters T, Ruan J, Amisaki M, Zebboudj A, Odgerel Z, Payne G, Derhovanessian E, Muller F, Rhee I, Yadav M, Dobrin A, Sadelain M, Luksza M, Cohen N, Tang L, Basturk O, Gonen M, Katz S, Do RK, Epstein AS, Momtaz P, Park W, Sugarman R, Varghese AM, Won E, Desai A, Wei AC, D'Angelica MI, Kingham TP, Mellman I, Merghoub T, Wolchok JD, Sahin U, Tureci O, Greenbaum BD, Jarnagin WR, Drebin J, O'Reilly EM, Balachandran VP. Personalized RNA neoantigen vaccines stimulate T cells in pancreatic cancer. Nature. 2023 Jun;618(7963):144-150. doi: 10.1038/s41586-023-06063-y. Epub 2023 May 10. PMID 37165196